CLINICAL TRIAL: NCT05471843
Title: A Single-Arm, Open-Label, Multicenter Phase 1/2 Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of BCL2 Inhibitor BGB-11417 in Patients With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: Study of BGB-11417 Monotherapy in Participants With Relapsed or Refractory Mantle Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BGB-11417-201; CTR20221815 (Other: ChinaDrugTrials); 2022-500687-35-00 (EU CTIS Number)
Record Dates: First submitted 2022-07-21; First posted 2022-07-25 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Mantle Cell Lymphoma; Refractory Mantle Cell Lymphoma (MCL); Relapsed Mantle Cell Lymphoma
Keywords: Mantle Cell Lymphoma; Lymphoma; MCL; Refractory MCL; Refractory Mantle Cell Lymphoma; Relapsed Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Participants will receive sonrotoclax
  Interventions: Drug: BGB-11417

INTERVENTIONS:
Drug: BGB-11417 — Administered orally
  Other Names: sonrotoclax

SUMMARY:
The study consists of two parts. Part 1 determines the safety and tolerability of BGB-11417 (sonrotoclax) monotherapy, the maximum tolerated dose, and the recommended Phase 2 dose of BGB-11417 monotherapy for relapsed or refractory mantle cell lymphoma. Part 2 evaluates efficacy of BGB-11417 monotherapy at the recommended Phase 2 dose with recommended ramp-up schedule from Part 1.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed diagnosis of MCL
2. Prior systemic treatments for MCL (at least one line of anti-cluster of differentiation 20 (anti-CD20) based immune or chemoimmunotherapy and at least one kind of covalent or non-covalent adequate Bruton Tyrosine Kinase (BTK) inhibitor).
3. Relapsed/refractory disease
4. Presence of measurable disease
5. Availability of archival tissue confirming diagnosis of MCL, or willing to undergo fresh tumor biopsy
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2.
7. Adequate organ function

Key Exclusion Criteria:

1. Known central nervous system involvement by lymphoma
2. Prior malignancy other than MCL within the past 3 years, except for curatively treated basal or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or localized Gleason score 6 prostate cancer.
3. Prior exposure to a BCL-2 inhibitor (eg, venetoclax/ABT-199).
4. Prior autologous stem cell transplant within the last 3 months; or prior autologous chimeric antigen receptor T-cell therapy within the last 3 months; or prior allogeneic stem cell transplant within the last 6 months or currently has an active graft-vs-host disease requiring the use of immunosuppressants.
5. Clinically significant cardiovascular disease.
6. Major surgery or significant injury ≤ 4 weeks prior to start of study treatment.
7. Active fungal, bacterial or viral infection requiring systemic treatment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number Of Participants Experiencing Dose-limiting Toxicities (DLTs) | Up to 1 Year
Part 1: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and adverse events leading to discontinuation. | Up to 5 Years
Part 1: Number of participants experiencing tumor lysis syndrome (TLS) relevant events | Up to 5 Years
Part 2: Overall Response Rate (ORR) as assessed by the Independent Review Committee (IRC) | Up to 4 Years
  Defined as the proportion of participants who achieved a complete response (CR), or partial response (PR) per the Lugano Classification

SECONDARY OUTCOMES:
Part 1: Single Dose Area Under the Plasma Concentration Time Curve (AUC) | Up to 2 Years
Part 1: Single Dose Maximum Observed Plasma Concentration (Cmax) | Up to 2 Years
Part 1: Single Dose Time to reach Cmax (Tmax) | Up to 2 Years
Part 1: Steady State Area Under the Plasma Concentration Time Curve (AUC) | Up to 2 Years
Part 1: Steady State Maximum Observed Plasma Concentration (Cmax) | Up to 2 Years
Part 1: Steady State Trough Plasma Concentration (CTrough) | Up to 2 Years
Part 1: Steady State Time to reach Cmax (Tmax) | Up to 2 Years
Overall Response Rate (ORR) as assessed by investigator | Up to 4 Years
  Defined as the proportion of participants who achieved a complete response (CR), or partial response (PR) per Lugano classification
Duration of Response (DOR) as assessed by investigator and IRC | Up to 4 Years
  DOR is defined as the time from the date of the first documented response (PR or better) after treatment initiation until the date of first documented disease progression or death due to any cause; whichever occurs first
Progression Free Survival (PFS) as assessed by investigator and IRC | Up to 4 Years
  PFS is defined as the time from the date of the first study dose until the date of first documented disease progression or death due to any cause, whichever occurs first.
Time to Response (TTR) as assessed by investigator and IRC | Up to 4 Years
  TTR is defined as the time from start of treatment to first documentation of response of Partial Response (PR) or better
Overall Survival (OS) | Up to 4 Years
  Defined as time from the start of treatment to the date of death due to any cause
Part 2: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and adverse events leading to discontinuation. | Up to 4 Years
Part 2: Number of participants with clinically significant changes from baseline in vital signs | Up to 4 Years
  Vital signs include blood pressure and pulse rate
Part 2: Number of participants with clinically significant changes from baseline in clinical laboratory values | Up to 4 Years
  Laboratory values include hematology, and clinical chemistry
Part 2: Number of Participants With Clinically Significant Physical Examination Findings | Up to 4 Years
  A Physical examination includes head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal and musculoskeletal systems
Part 2: Participant Reported Outcomes as measured by NFLymSI-18 | Up to 4 Years
  The National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy Lymphoma Cancer Symptom Index-18 (FLymSI-18) questionnaire contains 18 items, each of which utilizes a Likert scale with 5 possible responses ranging from 0 'Not at all' to 4 'Very much' and is divided into a total score.
Part 2: Participant Reported Outcomes as measured by EQ-5D-5L questionnaires | Up to 4 Years
  The EQ-5D-5L descriptive system assesses health in five dimensions (MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN / DISCOMFORT, ANXIETY / DEPRESSION), each of which has five levels of response (no problems, slight problems, moderate problems, severe problems, extreme problems/unable to). This part of the EQ-5D questionnaire provides a descriptive profile that can be used to generate a health state profile. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility. The second part of the questionnaire consists of a visual analogue scale (VAS) on which the participant rates his/her perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).

CONTACTS AND LOCATIONS:
Locations (104):
- United States (13):
  - University of Alabama At Birmingham Hospital, Birmingham, Alabama
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Des Moines Oncology Research Association, Des Moines, Iowa
  - Tulane Cancer Center, New Orleans, Louisiana
  - Luminis Health Anne Arundel Medical Center, Annapolis, Maryland
  - Maryland Oncology Hematology, Pa, Columbia, Maryland
  - University of Missouri Hospital, Ellis Fischel Cancer Center, Columbia, Missouri
  - Nebraska Cancer Specialists, Grand Island, Nebraska
  - Dartmouth Cancer Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Novant Health Hematology Charlotte, Charlotte, North Carolina
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
- Hospital Aleman, Buenos Aires, Argentina
- Belgium (4):
  - Az Sint Jan Brugge, Bruges
  - Universitair Ziekenhuis Gent, Ghent
  - University Hospitals Leuven, Leuven
  - AZ DELTA, Roeselare
- Brazil (11):
  - Hospital Erasto Gaertner, Curitiba
  - Hospital Mae de Deus, Porto Alegre
  - Hospital Das Clinicas Da Faculdade de Medicina de Ribeirao Preto Usp, Ribeirão Preto
  - Oncoclinicas Rio de Janeiro Sa, Rio de Janeiro
  - Instituto Americas Ensino, Pesquisa E Inovacao, Rio de Janeiro
  - Hospital Sao Rafael (Rede Dor), Salvador
  - Hospital Beneficencia Portuguesa de Sao Paulo, São Paulo
  - Instituto Dor de Pesquisa E Ensino Sao Paulo, São Paulo
  - Accamargo Cancer Center, São Paulo
  - Hcfmusp Servico de Hematologia, Hemoterapia E Terapia Celular, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- Qeii Health Science Center, Halifax, Nova Scotia, Canada
- China (32):
  - Anhui Provincial Cancer Hospital Aka West Branch of Anhui Province Hospital, Hefei, Anhui
  - China Japan Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital Medical University(Tongzhou), Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital Huifu Branch, Guangzhou, Guangdong
  - Jiangmen Central Hospital, Jiangmen, Guangdong
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Jiangxi Province Cancer Hospital, Nanchang, Jiangxi
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University Branch West Coast, Qingdao, Shandong
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Institute of Hematology and Hospital of Blood Disease, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Peoples Hospital of Kashgar, Kashgar, Xinjiang
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- France (6):
  - Centre Hospitalier Le Mans, Le Mans
  - Centre Hospitalier Universitaire Nantes Hotel Dieu, Nantes
  - Hopital Pitie Salpetriere Service Hematologie, Paris
  - Necker University Hospital, Paris
  - Chu Hopital Lyon Sud, PierreBenite
  - Chu Tours Hopital Bretonneau Service Pneumologie, Tours
- Germany (4):
  - Universitatsklinikum Koln, Innere Medizin I, Cologne
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Universitatsklinikum Essen (Aor), Essen
  - Universitatsklinikum Schleswig Holstein, Campus Kiel, Kiel
- Israel (6):
  - Assuta Ashdod Medical Center, Ashdod
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah En Karem Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Tel Aviv
  - Sourasky Tel Aviv Medical Center, Tel Aviv
- Italy (5):
  - Irccs Istituto Tumori Giovanni Paolo Ii, Bari
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia, Brescia
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori Irst, Meldola
  - Aou Maggiore Della Carita, Novara
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia McM Krakow, Krakow
  - Uniwersytecki Szpital Kliniczny Nr W Lublinie, Lublin
  - Narodowy Instytut Onkologii Im Marii Skodowskiej Curie Pastwowy Instytut Badawczy, Warsaw
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- Spain (3):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
- Turkey (Türkiye) (9):
  - Ankara University Medical Faculty, Ankara
  - Dr Abdurrahman Yurtaslan Oncology Teaching and Research Hospital, Ankara
  - Gazi University, Ankara
  - Ondokuz Mayis University Medicine Faculty Hospital, Atakum Samsun
  - Bagcilar Medipol Mega Hospital, Istanbul
  - Vkv American Hospital, Istanbul
  - Ege University Medical Faculty, Izmir
  - Erciyes University School of Medicine, Kayseri
  - Kocaeli Universitesi Tip Fakultesi, Kocaeli
- United Kingdom (4):
  - The Christie Hospital, Greater Manchester
  - Churchill Hospital Oxford University Hospital Nhs Trust, Headington
  - University College Hospital, London
  - Clatterbridge Cancer Centre, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes